CLINICAL TRIAL: NCT03764033
Title: A Novel Posttraumatic Stress Disorder Treatment for Veterans With Moral Injury
Acronym: IOK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D2946-R; I01RX004243 (NIH)
Record Dates: First submitted 2018-12-03; First posted 2018-12-04 (Actual); Results first posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Moral Injury
Keywords: Stress Disorders, Post-Traumatic; Moral Injury; Treatment
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: The investigators propose to conduct a multi-site, randomized, controlled trial to test the efficacy of an individual treatment for PTSD stemming from moral injury called IOK, compared to a present-centered therapy (PCT) control condition.
Who Masked: Outcomes Assessor
Masking Description: The clinical evaluators will be kept blind to treatment condition throughout the study period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Impact of Killing (IOK) (Experimental): Participants in this arm will receive 10 sessions (60-90 minutes) of a cognitive-behavioral moral injury treatment called IOK .
  Interventions: Behavioral: Impact of Killing (IOK)
- Present Centered Therapy (Active Comparator): Participants in this arm will receive 10 sessions (60-90 minutes) of a PTSD treatment that does not focus on trauma or cognitive restructuring, but rather the functional impact of trauma called Present Center Therapy (PCT)
  Interventions: Behavioral: Present Centered Therapy

INTERVENTIONS:
Behavioral: Impact of Killing (IOK) — Participants in this arm will receive 10 sessions (60-90 minutes) of a cognitive-behavioral moral injury treatment called IOK .
  Arms: Impact of Killing (IOK)
Behavioral: Present Centered Therapy — Participants in this arm will receive 10 sessions (60-90 minutes) of a PTSD treatment that does not focus on trauma or cognitive restructuring, but rather the functional impact of trauma called Present Center Therapy (PCT)
  Arms: Present Centered Therapy

SUMMARY:
The objective of this project is to test the efficacy of an individual treatment for post-traumatic stress disorder (PTSD) stemming from moral injury called Impact of Killing (IOK), compared to a present-centered therapy (PCT) control condition, and to determine the rehabilitative utility of IOK for Veterans with PTSD. The first aim is to test whether IOK can help improve psychosocial functioning for Veterans, as well as PTSD symptoms. The second aim is to determine whether IOK gains made by Veterans in treatment are durable, as measured by a six-month follow-up assessment. Veterans who kill in war are at increased risk for functional difficulties, PTSD, alcohol abuse, and suicide. Even after current PTSD psychotherapies, most Veterans continue to meet diagnostic criteria for PTSD, highlighting the need for expanding treatments for PTSD and functioning. IOK is a treatment that can be provided following existing PTSD treatments, filling a critical gap for Veterans with moral injury who continue to suffer from mental health symptoms and functional difficulties.

DETAILED DESCRIPTION:
Post-traumatic stress disorder (PTSD) is now the most common mental health diagnosis among the youngest generation of Veterans receiving treatment from the Veterans Health Administration (VHA), necessitating the need for diverse types of targeted care. Although there are two evidence-based psychotherapies (EBP) for PTSD, the vast majority of combat Veterans who receive these treatments still meet diagnostic criteria for PTSD and their functioning continues to be impacted. Furthermore, Veterans that have experienced trauma related to killing have high rates of suicide and more severe PTSD symptoms. Although there have been few studies examining predictors of poor outcomes in EBPs, one area that has recently begun to receive growing attention is moral injury. A recent study found that PTSD and moral injury were distinct constructs with unique signs and symptoms, and preliminary evidence indicates that the feelings of guilt and anger that characterize moral injury associated with trauma such as killing in war may contribute to worsening symptoms over the course of existing treatments. Although PTSD may be one manifestation of psychological trauma related to killing, conceptualization of the impact of killing requires a broader framework. The emerging concept of moral injury offers an alternative context to better understand the many possible outcomes of exposure to killing. For these reasons, the development of targeted moral injury interventions is critical. The investigators designed and received VA funding to conduct a pilot randomized controlled trial (RCT) of the Impact of Killing (IOK) treatment, which can be seamlessly added as a standalone treatment following existing EBPs for PTSD. IOK focuses on key themes including physiology of killing responses, moral injury, self-forgiveness, and improved post-deployment reintegration. The treatment was designed to fit well into already existing systems of care and has been shown to improve functioning, PTSD symptoms, and general psychiatric symptoms following EBP. Whereas the IOK RCT pilot was initially conducted at the San Francisco VA Healthcare System, the investigators' goal is to conduct a fully-powered, multi-site efficacy trial at two regionally-diverse sites with a larger sample size and active control condition. Consequently, the objective of this project is to test the efficacy of an individual treatment for PTSD stemming from moral injury called IOK, compared to a present-centered therapy (PCT) control condition, and to determine the rehabilitative utility of IOK for Veterans seeking treatment for PTSD. The primary outcome is psychosocial functioning. The target population is Veterans who have initiated or completed Cognitive Processing Therapy or Prolonged Exposure Therapy, two EBPs for PTSD, and continue to have PTSD symptoms and moral injury related to killing. Veterans will be randomly assigned to receive either: 1) IOK (10 individual therapy sessions lasting 60-90 minutes) or 2) PCT (sessions of equal duration to IOK). The first aim is to test the efficacy of IOK through measures of psychosocial functioning (primary outcome) and PTSD severity (secondary outcome). The second aim is to determine whether IOK gains made by Veterans are durable. If the aims of this grant are achieved, the investigators will be able to have a moral injury intervention following EBP that can be seamlessly integrated into existing care for one of the most commonly occurring mental health problems in Veterans. Furthermore, suicide is a national priority for VHA, and expanding treatment for PTSD and moral injury has the potential to decrease suicide and improve functioning in Veterans. Finally, IOK offers skills and ways of understanding warzone experiences that can be mastered and can continue to be implemented by Veterans over time.

ELIGIBILITY:
Inclusion Criteria:

* Veterans 18-82 years of age
* Veterans who meet Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for Post-traumatic Stress Disorder (PTSD) or score 23 or higher on the Clinician-Administered PTSD Scale for DSM-5 (CAPS) screening interview.
* Veterans who endorsed killing or being responsible for the death of another in a war zone and report continued distress regarding these events

  * Distress will be operationalized by a positive response to one or more of the nine self-directed moral injury items on the Expressions of Moral Injury Scale-Military Version (EMIS-M) or item #4 on the Moral Injury Events Scale (MIES)
* Veterans who have initiated or completed an evidence-based treatment for PTSD, such as Cognitive Processing Therapy (CPT) or Prolonged Exposure (PE)
* If receiving CPT or PE, Veterans must complete treatment and wait two weeks prior to screening
* If receiving prescription medication for PTSD, Veterans must be one month stable on medication and not make any changes to medication during the course of the active treatment phase of the study

Exclusion Criteria:

* Veterans with current or lifetime diagnosis of a psychotic disorder or current untreated/unmanaged mania.
* Veterans with recent suicidal or homicidal behaviors (chronic suicidal ideation is not exclusionary)
* Veterans with recent psychiatric hospitalizations
* Veterans with moderate or severe alcohol or drug dependence within the past three months
* Veterans receiving individual therapy for PTSD or those planning to start skills-based or trauma-focused group psychotherapy will be excluded

  * However, these Veterans will be offered the opportunity to be screened again after completion of individual PTSD therapy or once they are three months stable in group treatment, with no plans to discontinue this treatment

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shira Maguen, PhD, Principal Investigator — San Francisco VA Medical Center, San Francisco, CA
Locations (3):
- United States (3):
  - San Francisco VA Medical Center, San Francisco, CA, San Francisco, California
  - James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Veterans were recruited from 8/12/2019 to 11/30/2024 through direct mailings, advertisements, referrals from VA providers and other VA research studies. Screening procedures comprised a brief phone pre-screener, informed consent , and a diagnostic clinical interview. A total of 100 Veterans completed all screening procedures, were eligible for the study, completed a baseline self-report questionnaire of outcome measures, and were randomly assigned to a treatment condition.
Period: Treatment Phase
Arm/Group | Impact of Killing (IOK) | Present Centered Therapy
Started (Enrolled & Randomized to Treatment Condition) | 49 | 51
Completed (Completed Study Treatment) | 41 | 47
Not Completed | 8 | 4
Not completed — Withdrawal by Subject | 8 | 3
Not completed — Withdrawn by PI due to frequent no-shows and cancellations of study appointments. | 0 | 1
Period: Six Month Follow-Up
Arm/Group | Impact of Killing (IOK) | Present Centered Therapy
Started (Completed Treatment and Sent Follow-up Questionnaires) | 41 | 47
Completed (Completed Six-Month Follow-up Questionnaires) | 41 | 42
Not Completed | 0 | 5
Not completed — Lost to Follow-up | 0 | 5

BASELINE CHARACTERISTICS:
Population: Participants that passed all screening procedures and were eligible for treatment randomization & enrollment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Impact of Killing (IOK) | Present Centered Therapy | Total
Number analyzed (Participants) | 49 | 51 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.0 (14.5) | 46.8 (12.9) | 48.4 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 48 | 50 | 98
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 11 | 19
  Not Hispanic or Latino | 41 | 40 | 81
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 13 | 25
  White | 34 | 34 | 68
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: World Health Organization Quality of Life-BREF
Description: A widely-validated, 26-item measure on a 5 point scale that assesses functioning in physical health, psychological health, social relationships, and environment, with higher scores indicating greater health in each domain. Each item is scored from 1-5, and a total raw score is calculated by summing all items (26-130). The total score is calculated by transforming the raw score to a 0-100 scale, with higher scores representing better quality of life.
Time Frame: Change from baseline (Week 0) and post-treatment (Week 11)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Impact of Killing (IOK) | Present Centered Therapy
Number analyzed (Participants) | 49 | 51
score on a scale | 53.35 (2.03) | 52.39 (1.94)
Statistical Analysis 1: Comparison: Impact of Killing (IOK) vs Present Centered Therapy; Test type: Superiority; p = 0.729, Mixed Models Analysis — The threshold for statistical significance was p=.05; Mean Difference (Net) = 0.78, 95% CI 2-sided [-3.66 to 5.24], Standard Error of Mean 2.27

2. Primary Outcome: World Health Organization Quality of Life-BREF
Description: as for outcome 1
Time Frame: Change from post-treatment (Week 11) to 6 month follow-up (6 months after post-treatment)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Impact of Killing (IOK) | Present Centered Therapy
Number analyzed (Participants) | 41 | 42
score on a scale | 50.86 (2.03) | 50.62 (1.99)
Statistical Analysis 1: Comparison: Impact of Killing (IOK) vs Present Centered Therapy; Test type: Superiority; p = 0.975, Mixed Models Analysis — The threshold for statistical significance was p=.05; Mean Difference (Net) = 0.07, 95% CI 2-sided [-4.46 to 4.61], Standard Error of Mean 2.31

3. Secondary Outcome: Clinician Administered PTSD Scale for DSM-5 (CAPS-5)
Description: This measure is used to identify DSM-5 criteria for PTSD. CAPS-5 provides both a dimensional and categorical measure of current PTSD and the frequency and intensity of PTSD-related symptoms. Score range from 0-80 with lower score representing fewer PTSD symptoms.
Time Frame: Change from baseline (Week 0) and post-treatment (Week 11)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Impact of Killing (IOK) | Present Centered Therapy
Number analyzed (Participants) | 49 | 51
score on a scale | 25.79 (1.82) | 26.03 (1.73)
Statistical Analysis 1: Comparison: Impact of Killing (IOK) vs Present Centered Therapy; Test type: Superiority; p = 0.831, Mixed Models Analysis — The threshold for statistical significance was p=.05; Mean Difference (Net) = -0.52, 95% CI 2-sided [-5.27 to 4.24], Standard Error of Mean 2.43

4. Other Pre Specified Outcome: PTSD Checklist for DSM-5 (PCL-5)
Description: A 20-item measure that assesses PTSD symptom severity using a 5-point rating scale. The PCL-5 items correspond to the DSM-5 symptoms for PTSD. Total severity can range from 0 to 80. Higher scores indicate greater severity of PTSD symptoms.
Time Frame: Change from baseline (Week 0) and post-treatment (Week 11)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Impact of Killing (IOK) | Present Centered Therapy
Number analyzed (Participants) | 49 | 51
score on a scale | 37.31 (2.23) | 42.9 (2.14)
Statistical Analysis 1: Comparison: Impact of Killing (IOK) vs Present Centered Therapy; Test type: Superiority; p = 0.006, Mixed Models Analysis — The threshold for statistical significance was p=.05; Mean Difference (Net) = -6.59, 95% CI 2-sided [-11.31 to -1.87], Standard Error of Mean 2.42

5. Other Pre Specified Outcome: PTSD Checklist for DSM-5 (PCL-5)
Description: as for outcome 4
Time Frame: Change from post-treatment (Week 11) to 6 month follow-up (6 months after post-treatment)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Impact of Killing (IOK) | Present Centered Therapy
Number analyzed (Participants) | 41 | 42
score on a scale | 36.77 (2.23) | 42.35 (2.19)
Statistical Analysis 1: Comparison: Impact of Killing (IOK) vs Present Centered Therapy; Test type: Superiority; p = 0.008, Mixed Models Analysis — The threshold for statistical significance was p=.05; Mean Difference (Net) = -6.54, 95% CI 2-sided [-11.34 to -1.74], Standard Error of Mean 2.44

6. Other Pre Specified Outcome: Brief Symptom Inventory (BSI)
Description: A 53-item measure, using a 5-point Likert scale, in which participants rate the extent to which they have been bothered in the past week by various mental health symptoms (e.g., depression, anxiety, hostility, psychoticism, paranoid ideation, etc.). The BSI measures global psychological distress, with scores ranging from 0-53. Higher scores represent more severe psychiatric symptoms.
Time Frame: Change from baseline (Week 0) and post-treatment (Week 11)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Impact of Killing (IOK) | Present Centered Therapy
Number analyzed (Participants) | 49 | 51
score on a scale | 1.11 (0.11) | 1.35 (0.10)
Statistical Analysis 1: Comparison: Impact of Killing (IOK) vs Present Centered Therapy; Test type: Superiority; p = 0.066, Mixed Models Analysis — The threshold for statistical significance was p=.05; Mean Difference (Net) = -0.18, 95% CI 2-sided [-0.37 to 0.01], Standard Error of Mean 0.11

7. Other Pre Specified Outcome: Trauma-related Guilt Inventory (TRGI)
Description: A 32-item measure, using a 5-point Likert scale, assessing the emotional and cognitive aspects of guilt associated with a specified traumatic event (e.g., combat experience, car accident, physical or sexual abuse, or sudden death of a loved one). The TRGI has main scales representing guilt, distress and guilt cognitions. Scores represent the average for items in the scale and range from 0-4, with higher scores representing greater guilt/distress.
Time Frame: Change from baseline (Week 0) and post-treatment (Week 11)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Impact of Killing (IOK) | Present Centered Therapy
Number analyzed (Participants) | 49 | 51
score on a scale | 2.01 (0.15) | 2.18 (0.14)
Statistical Analysis 1: Comparison: Impact of Killing (IOK) vs Present Centered Therapy; Test type: Superiority; p = 0.043, Mixed Models Analysis — The threshold for statistical significance was p=.05; Mean Difference (Net) = -0.35, 95% CI 2-sided [-0.69 to -0.01], Standard Error of Mean 0.17

8. Other Pre Specified Outcome: Brief Symptom Inventory (BSI)
Description: as for outcome 6
Time Frame: Change from post-treatment (Week 11) to 6 month follow-up (6 months after post-treatment)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Impact of Killing (IOK) | Present Centered Therapy
Number analyzed (Participants) | 41 | 42
score on a scale | 1.15 (0.11) | 1.45 (0.10)
Statistical Analysis 1: Comparison: Impact of Killing (IOK) vs Present Centered Therapy; Test type: Superiority; p = 0.016, Mixed Models Analysis — The threshold for statistical significance was p=.05; Mean Difference (Net) = -.24, 95% CI 2-sided [-0.43 to -0.04], Standard Error of Mean 0.10

9. Other Pre Specified Outcome: Trauma-related Guilt Inventory (TRGI)
Description: A 32-item measure, using a 5-point Likert scale, assessing the emotional and cognitive aspects of guilt associated with a specified traumatic event (e.g., combat experience, car accident, physical or sexual abuse, or sudden death of a loved one). The TRGI has main scales representing guilt, distress and guilt cognitions. Scores represent the average for items in the scale and range from 0-4, with higher scores representing more guilt/distress.
Time Frame: Change from post-treatment (Week 11) to 6 month follow-up (6 months after post-treatment)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Impact of Killing (IOK) | Present Centered Therapy
Number analyzed (Participants) | 41 | 42
score on a scale | 1.79 (0.15) | 2.00 (0.15)
Statistical Analysis 1: Comparison: Impact of Killing (IOK) vs Present Centered Therapy; Test type: Superiority; p = 0.028, Mixed Models Analysis — The threshold for statistical significance was p=.05; Mean Difference (Net) = -0.39, 95% CI 2-sided [-0.74 to -0.04], Standard Error of Mean 0.18

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for participants during the treatment phase of the study, from baseline (Week 0) to the post-treatment diagnostic interview (Week 11)
Arm/Group | Impact of Killing (IOK) | Present Centered Therapy
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/51
Other Adverse Events (participants affected / at risk) | 0/49 | 1/51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Impact of Killing (IOK) (N=49) | Present Centered Therapy (N=51)
Drug Relapse (Psychiatric disorders) | 0 (0) | 1 (1) — Individual with prior history of a substance use disorder relapsed during treatment and withdrew from the study to focus on substance use therapy.

LIMITATIONS AND CAVEATS:
The study began prior to the Covid-19 pandemic. Three participants completed all data collection procedures and treatment in-person before the pandemic lockdown. The remaining participants completed some (n=5) or all (n=92) study procedures during the pandemic, through video or in-person appointments (as restrictions were lifted) and paper or electronic data collection methods.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-10-23): https://cdn.clinicaltrials.gov/large-docs/33/NCT03764033/Prot_SAP_000.pdf